CLINICAL TRIAL: NCT02874872
Title: Building a Novel Antibiotic Stewardship Intervention for Nursing Homes
Acronym: OASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0274
Record Dates: First submitted 2016-08-09; First posted 2016-08-22 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Antibiotics
Keywords: Nursing homes; Antibiotic Stewardship; Antibiotic Resistance
MeSH Terms: interventions — poly(divinyl-co-N-vinylpyrrolidinone)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OASIS Collaborative (Experimental): The nursing homes in this arm will receive facilitated implementation of two tools aimed at minimizing unnecessary antibiotic use. Facilitated implementation includes coaching of the nursing home staff on use of the tools. In addition, nursing home management will be coached on how to monitor implementation fidelity, antibiotic utilization, and consequences to over- and under-utilization of antibiotics as feedback on the effectiveness of the intervention. Finally, nursing home management will receive coaching on how to develop and implement a sustain plan for the OASIS intervention.
  Interventions: Behavioral: OASIS Collaborative
- Control (No Intervention): The nursing homes in this arm will continue care as usual, with no tools or facilitated implementation.

INTERVENTIONS:
Behavioral: OASIS Collaborative — OASIS (Optimizing Antibiotic Stewardship in Skilled Nursing Facilities) is a system redesign of skilled nursing facility work systems
  Other Names: OASIS
  Arms: OASIS Collaborative

SUMMARY:
The OASIS Collaborative is an organizational intervention aimed at reducing unnecessary antibiotic use in skilled nursing facilities. The first target of intervention is the tasks carried out by nursing staff after a change in condition and after an antibiotic prescription is initiated. The second target are the management staff who provide feedback to staff. The third target are the administrators who identify and overcome organizational barriers to implementation.

In this study, we will implement two tools that are intended to minimize unnecessary antibiotic use in skilled nursing facilities. The first tool helps skilled nursing facility staff assess risk and communicate with prescribers when residents experience a change in health status that may result in the use of antibiotics. The second tool is used after an antibiotic is prescribed; the tool streamlines reassessment of the patient, and provides prescribers the opportunity to consider stopping unnecessary antibiotic prescriptions, narrowing the spectrum of antibiotic therapy, or shortening the duration of antibiotic therapy.

ELIGIBILITY:
This is an organizational intervention. Outcomes will be evaluated at the population-level by facility.

Nursing home residents:

Inclusion Criteria:

* Any nursing home resident who has received antibiotic therapy in any of the 12 participating nursing home facilities.

Exclusion Criteria:

* Nursing home residents who have not received antibiotic therapy in any of the 12 participating nursing home facilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2942 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Days of Antibiotic Therapy (DOT)/1000 resident days | up to 12 months
  Utilization of antibiotics initiated in the nursing home, defined as the number of days a nursing home resident receives antibiotic therapy.
  This measure includes antibiotic courses initiated 1) in the nursing home or 2) Emergency Department, if the resident returned to the nursing home without intercurrent hospitalization. This measure excludes antibiotic courses started during a hospital stay and continued in the nursing home after discharge.
Proportion of Antibiotic Starts meeting Loeb Criteria | up to 12 months
  Defined as the proportion of antibiotic courses started in the nursing home or Emergency department that satisfy the Loeb minimum criteria for initiation of antibiotics.
  This measure includes antibiotic courses initiated 1) in the nursing home or 2) Emergency Department, if the resident returned to the nursing home without intercurrent hospitalization. This measure excludes antibiotic courses started during a hospital stay and continued in the nursing home after discharge.

SECONDARY OUTCOMES:
Incidence of antibiotic starts/1000 resident days | up to 12 months pre-implementation and up to 12 months post-implementation
  Defined as the number of antibiotic courses started per 1000 resident days.
  This measure includes antibiotic courses initiated 1) in the nursing home or 2) Emergency Department, if the resident returned to the nursing home without intercurrent hospitalization. This measure excludes antibiotic courses started during a hospital stay and continued in the nursing home after discharge.
Fluoroquinolone Days of Therapy (FQD)/1000 resident days | up to 12 months pre-implementation and up to 12 months post-implementation
  Defined as the number of days a nursing home resident receives fluoroquinolone therapy.
  This measure includes antibiotic courses initiated 1) in the nursing home or 2) Emergency Department, if the resident returned to the nursing home without intercurrent hospitalization. This measure excludes antibiotic courses started during a hospital stay and continued in the nursing home after discharge.
Incidence of C.diff infection/1000 resident days | up to 12 months pre-implementation and up to 12 months post-implementation
  Defined as the number of positive C. difficile tests per 1000 resident days
Fluoroquinolone resistance | up to 12 months pre-implementation and up to 12 months post-implementation
  Defined as the proportion of urine cultures that grow bacteria that are resistant to fluoroquinolone antibiotics.
Positive Enterococcus species | up to 12 months pre-implementation and up to 12 months post-implementation
  Defined as the proportion of urine cultures that grow Enterococcus species
Positive Candida species | up to 12 months pre-implementation and up to 12 months post-implementation
  Defined as the proportion of urine cultures that grow Candida species

OTHER OUTCOMES:
Incidence of nursing home deaths/1000 resident days | up to 12 months pre-implementation and up to 12 months post-implementation
  Includes deaths that occur in 1) the nursing home or 2) the hospital if a resident's bed is kept on hold at the nursing home.
Incidence of unplanned transfers/1000 resident days | up to 12 months pre-implementation and up to 12 months post-implementation
  Includes unplanned transfers to 1) the hospital or 2) the emergency room that do not result in hospitalization. This measure excludes planned transfers (e.g., physician clinic visits) or hospitalizations (e.g., for a planned surgical procedure or other therapy).
Combined deaths and unplanned transfers/1000 resident days | up to 12 months pre-implementation and up to 12 months post-implementation
  Defined as the sum of deaths and unplanned transfers, as defined above.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Crnich, MD, PhD, Principal Investigator — University of Wisconsin-Madison, School of Medicine and Public Health; James H Ford II, PhD, Principal Investigator — University of Wisconsin-Madison, College of Engineering; David A Nace, MD, MPH, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: No